CLINICAL TRIAL: NCT03555370
Title: RCT of Vestibular Treatment in Adolescents Following Sport Related Concussion
Brief Title: Vestibular Treatment in Adolescents Following Sport Related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Associate Professor, Dept of Orthopaedic Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO18020291
Record Dates: First submitted 2018-05-11; First posted 2018-06-13 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Vestibular Disorder
Keywords: adolescent; concussion
MeSH Terms: conditions — Vestibular Diseases; Brain Concussion | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (Experimental): Standard of Care:
  The standard of care protocol consists of standardized in office and at home behavioral management to include sleep, hydration, nutrition, and stress management interventions. Participants will also be assigned physical activity that they will complete during their visits and at home. Physical activity for the standard of care group will include 15 minutes of flexibility/range of motion exercises, and 10 minutes of aerobic-based daily physical activity (e.g.,walking, stationary cycle).
  Interventions: Behavioral: Standard of Care
- Vestibular Exercise Intervention Group (Experimental): The vestibular group will complete the behavioral management activities described above, as well as prescribed in-office and at home vestibular exercises from each of four groups: 1) gaze stability training (i.e., integrated eye and head movements on fixed target), 2) visual motion training (i.e., integrated eye and head movements with busy visual background), 3) standing balance (i.e., standing in different stances), and 4) dynamic gait (i.e., walking with head turns). Participants will be prescribed to one of four levels of these four exercise groups based on presentation of symptoms/impairment as indicated on the VOMS. Progression through the four levels will be based on symptom tolerance and successful completion of all exercises at the current level.
  Interventions: Behavioral: Vestibular Exercise Intervention

INTERVENTIONS:
Behavioral: Vestibular Exercise Intervention — The vestibular exercise intervention group will complete behavioral management activities, and prescribed in--office/at home vestibular exercises from four groups: 1) gaze stability training (integrated eye and head movements on fixed target), 2) visual motion training (integrated eye and head movements on moving target), 3) standing balance (standing with eyes closed in different stances), and 4) dynamic gait (walking with head turns and eye movements). Participants will be prescribed to one of four levels of these exercise groups based on presentation of symptoms/impairment as indicated on VOMS. Progression through the levels will be based on symptom tolerance and successful completion of all exercises at the current level.
  Arms: Vestibular Exercise Intervention Group
Behavioral: Standard of Care — The standard of care consists of standardized in office/at home behavioral management including sleep, hydration, nutrition, and stress management interventions.
  Arms: Standard of Care Group

SUMMARY:
Each year, nearly 2 million children and adolescents have a sport-related concussion (SRC) in the U.S., but 57% of them do not receive appropriate clinical care following their injury. These injuries involve a wide range of symptoms including headache, dizziness, and sleep problems; and cognitive, emotional, visual, and vestibular impairment. The investigators have developed a clinical treatment model for SRC that addresses the heterogeneity of this injury using different clinical subtypes or profiles that inform precision interventions. To date, the investigators have identified cognitive, anxiety/mood, post-traumatic migraine, cervical, oculomotor, and vestibular clinical profiles. Patients with vestibular clinical profiles- involving dizziness, environmental sensitivity, and imbalance- are common (60-65% of concussions), and have worse outcomes and longer recovery following SRC. Consequently, the investigators have developed and applied precision vestibular treatments that can be matched to specific impairments and symptoms to actively treat patients with vestibular clinic profiles.

DETAILED DESCRIPTION:
To determine using a RCT design the effectiveness of standard of care behavioral management (i.e., sleep, walking, nutrition, stress management) to standard of care behavioral management (i.e., sleep, walking, nutrition, stress management) (STANDARD OF CARE) plus vestibular exercises (i.e., balance, eye-head movements, and dynamic walking exercises) (VESTIBULAR) for reducing recovery time, symptoms, and vestibular (balance, eye-head movements) and cognitive (e.g., memory, processing speed) impairment in adolescent patients with vestibular clinical profiles following sport--related concussion (SRC).

ELIGIBILITY:
Inclusion Criteria:

* Must be 12-18 years of age.
* Must be diagnosed with a sport-related concussion within the last 3-10 days.
* Must be identified by UPMC Sports Medicine clinicians as having clinical presentation of a vestibular profile of concussion.
* Must report an increase of +2 of symptom provocation on VOMS (from baseline symptom report) on either VOR or VMS measurements during VOMS assessment.

Exclusion Criteria:

* More than 3 concussions including presenting injury;
* Current history or pre-existing vestibular disorder;
* Current orthopaedic injury;
* History of brain surgery or TBI (based on Glasgow Coma Scale of <13);
* History of substance abuse;
* History of neurological disorder (seizure disorder, epilepsy, brain tumors or malformations);
* Current concussion is non-sport related.

The above exclusion factors are known to influence recovery and thus if any one exclusion criterion is met, the athlete will be unable to participate in the current study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Change in VOMS Scores (Vestibular Ocular Motor Screening) from Baseline to 4 Week/Visit 2 | Measures will be conducted at enrollment (within 10 days of injury) and at 2 weeks (+ or - 5 days) and 4 weeks (+ or - 5 days) following treatment.
  The VOMS assesses vestibular and ocular motor impairment via patient-reported symptom provocation brief assessments in 7 components: 1) smooth pursuits; 2, 3) horizontal and vertical saccades; 4) near point convergence (NPC); 5, 6) horizontal and vertical vestibular ocular reflex (VOR), and 7) visual motion sensitivity (VMS). Patients rate changes in headache, dizziness, nausea, and fogginess symptoms compared to immediate pre-assessment state on a scale of 0 (no symptoms) to 10 (severe symptoms) following each VOMS assessment to determine if each assessment provokes symptoms. Convergence is assessed by both symptom report and objective measurement of NPC distance, values are averaged across 3 trials. The VOMS takes approximately 5 min to administer.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Kontos, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UMPC Sports Medicine Concussion Research Program, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryan MA, Rowhani-Rahbar A, Comstock RD, Rivara F; Seattle Sports Concussion Research Collaborative. Sports- and Recreation-Related Concussions in US Youth. Pediatrics. 2016 Jul;138(1):e20154635. doi: 10.1542/peds.2015-4635. Epub 2016 Jun 20. PMID 27325635
- [Background] O'Kane JW, Schiff MA. Concerns about concussion rates in female youth soccer-reply. JAMA Pediatr. 2014 Oct;168(10):968. doi: 10.1001/jamapediatrics.2014.780. No abstract available. PMID 25285866
- [Background] Collins MW, Kontos AP, Okonkwo DO, Almquist J, Bailes J, Barisa M, Bazarian J, Bloom OJ, Brody DL, Cantu R, Cardenas J, Clugston J, Cohen R, Echemendia R, Elbin RJ, Ellenbogen R, Fonseca J, Gioia G, Guskiewicz K, Heyer R, Hotz G, Iverson GL, Jordan B, Manley G, Maroon J, McAllister T, McCrea M, Mucha A, Pieroth E, Podell K, Pombo M, Shetty T, Sills A, Solomon G, Thomas DG, Valovich McLeod TC, Yates T, Zafonte R. Statements of Agreement From the Targeted Evaluation and Active Management (TEAM) Approaches to Treating Concussion Meeting Held in Pittsburgh, October 15-16, 2015. Neurosurgery. 2016 Dec;79(6):912-929. doi: 10.1227/NEU.0000000000001447. PMID 27741219
- [Background] Mucha A, Collins MW, Elbin RJ, Furman JM, Troutman-Enseki C, DeWolf RM, Marchetti G, Kontos AP. A Brief Vestibular/Ocular Motor Screening (VOMS) assessment to evaluate concussions: preliminary findings. Am J Sports Med. 2014 Oct;42(10):2479-86. doi: 10.1177/0363546514543775. Epub 2014 Aug 8. PMID 25106780
- [Background] Collins MW, Kontos AP, Reynolds E, Murawski CD, Fu FH. A comprehensive, targeted approach to the clinical care of athletes following sport-related concussion. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):235-46. doi: 10.1007/s00167-013-2791-6. Epub 2013 Dec 12. PMID 24337463
- [Derived] Kontos AP, Eagle SR, Mucha A, Kochick V, Reichard J, Moldolvan C, Holland CL, Blaney NA, Collins MW. A Randomized Controlled Trial of Precision Vestibular Rehabilitation in Adolescents following Concussion: Preliminary Findings. J Pediatr. 2021 Dec;239:193-199. doi: 10.1016/j.jpeds.2021.08.032. Epub 2021 Aug 25. PMID 34450120